CLINICAL TRIAL: NCT02376218
Title: Post-lobectomy Use of Glucose for Pleurodesis and Air-leak Cessation. A Feasibility Trial.
Acronym: PLUG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Eric Frechette, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105807
Record Dates: First submitted 2015-02-20; First posted 2015-03-03 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Pulmonary Surgical Procedures

ARMS (1):
- Hypertonic 50% dextrose pleurodesis (Experimental)
  Interventions: Drug: Hypertonic 50% dextrose pleurodesis

INTERVENTIONS:
Drug: Hypertonic 50% dextrose pleurodesis — Intrapleural administration of 180ml of hypertonic dextrose solution.

SUMMARY:
It is common practice to leave a chest drainage catheter after lung surgical resections to manage air leaks. The air leakage will usually stop in the initial postoperative days, but in a few patients, it will last for a longer period of time, preventing the removal of the chest tube that can lead to patient discomfort, increased likelihood to develop postoperative complications and longer length of hospital stay. Pleurodesis is an effective method to address postoperative air leak which consists in injecting an irritating solution into the chest cavity. This is not performed regularly after lung resections for different reasons including associated pain, costs, and fear of infections. Pleurodesis with hyperosmolar glucose solution have been used for years with good results in some Asian countries because of its simplicity and low cost. Its effectiveness for pleurodesis has been reported in cases of spontaneous pneumothorax and chylothorax, but its efficiency to stop air leaks in the postoperative period remains to be defined.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older at the time of surgery
* Having undergone a simple lung lobectomy for malignancy, primary or metastatic
* Procedure performed through thoracotomy, sternotomy or video-assisted thoracic surgery (VATS), and associated or not to mediastinoscopy, staging thoracoscopy, mediastinal lymph nodes sampling or mediastinal lymph nodes dissection
* Normally recovery after a surgery performed between 12 and 24 hours earlier

Exclusion Criteria:

* High amount of liquid drainage from chest tube (>500 cc in the last 8 hours)
* Minimal air leak (<20 cc/min in one of the last 4 hours)
* Large air leak (>500 cc/min in one of the last 4 hours)
* History of previous ipsilateral thoracotomy, lung resection, rib fracture, chest trauma, or lung/thoracic infection
* Diabetes or hyperglycemia
* Immunity disorders
* Allergy to local anaesthetics
* Hemodynamic instability
* Need for respiratory support
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Air leak cessation | 48 hours after time of initial injection of 50% glucose solution
  air leak <20 cc/min for 4 hours or more

SECONDARY OUTCOMES:
Time to air leak cessation | 30-day post-operative period
Time to chest tube removal | 30-day post-operative period
Length of hospitalization | 30-day post-operative period
Postoperative complications | 30-day post-operative period
  number of participants with one of the following: o Hyperglycemia o De novo atrial fibrillation o Pneumonia o Empyema o Thromboembolic disorders o Confusion o Need for discharge with chest tube o Recurrent pneumothorax o Need for chest tube reinsertion o Death

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada